CLINICAL TRIAL: NCT04249817
Title: Keeping Stable Inflammatory Arthritis Patients in Their Communities With the Advanced Clinician Practitioner in Arthritis Care (ACPAC)
Brief Title: Keeping Stable Inflammatory Arthritis Patients in Their Communities With the Advanced Clinician Practitioner in Arthritis Care
Acronym: ACPAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Usual care was no longer possible with COVID19 and we no longer had a control for this study.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Initiative for Outcomes in Rheumatology Care (Other)
Responsible Party: Principal Investigator, Dr. Mary Bell, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 238-2019
Record Dates: First submitted 2019-09-17; First posted 2020-01-31 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video conferencing with extended role practitioner (Experimental): Participant goes to Ontario Telemedicine site for follow-up. At site, participant will get a physical assessment by an extended role practitioner and then will connect to their rheumatologist by videoconferencing for completion of follow-up.
  Interventions: Other: Video Conferencing with Exteneded Role Practitioner (VC-ERP)
- Usual care (No Intervention): Participant goes to their rheumatologist's clinic for follow-up, including physical assessment by their rheumatologist, as they would normally.

INTERVENTIONS:
Other: Video Conferencing with Exteneded Role Practitioner (VC-ERP) — Participant goes to Ontario Telemedicine site for follow-up. At site, participant will get a physical assessment by an extended role practitioner and then will connect to their rheumatologist by videoconferencing for completion of follow-up.
  Arms: Video conferencing with extended role practitioner

SUMMARY:
In Ontario, rheumatology services are in short supply. Many people with inflammatory arthritis (IA) are traveling long distances for care and face geographical/ financial challenges in so doing. Travel burden may be decreased and satisfaction with care improved by integrating existing health care resources. A few rheumatologists in Ontario have adopted a video conferencing (VC) model for follow-up of stable IA patients using the Ontario Telemedicine Network (OTN) with Extended Role Practitioners (ERPs) doing on-site assessments. Anecdotal evidence suggests this model benefits both patient and rheumatologist. We will determine how people with stable well-controlled IA, living more than 100 km round-trip from the rheumatology clinic, perceive quality of life before, during and after VC with ERP follow-up visits compared to usual care. Disease activity, functional status, medication adherence, patient satisfaction, and barriers to care will also be measured.

DETAILED DESCRIPTION:
Rationale: To determine, using a mixed-methods design, the impact of a rheumatology appointment via video conferencing combined with on-site pre-assessment by an Advance Clinician Practioner in Arthritis Care (ACPAC)-trained ERP compared to usual in-clinic care during a one-year period of follow-up for a cohort of persons with stable, well-controlled inflammatory arthritis residing in areas of low rheumatology supply.

Research Questions: For people with stable IA residing in areas of low rheumatology supply, is it feasible to provide follow-up to people with stable, well-controlled IA using videoconferencing and an assessment by an extended role practitioner? Does VC with ERP pre-assessment change quality of life and barriers to care perceived by people with stable, well-controlled IA?

Methods: Mixed-methods design. Randomized controlled trial with 2 groups: VC with ERP (VC-ERP) and usual care (UC). Pre- and Post-trial Interviews. Study procedures will be as follows:

1. Pre-trial Interview - 15 minute telephone interview that will be audio taped. Will take place no more than one month before baseline study visit. Participant will be asked about experience traveling to rheumatologist and barriers to receiving care closer to home.
2. Baseline visit - This visit will be a regularly scheduled appointment with the participant's rheumatologist. The participant will complete a package of four questionnaires and the rheumatologist will assess disease activity.
3. Randomization - after completion of the baseline visit, participants will be randomized either to VC-ERP or UC.
4. Follow-up Visits - There will be three follow-up visits 6, 12, and 13 months after the baseline study visit. Participants assigned to UC will be seen by their rheumatologist at the clinic as usual for all visits. At each visit, the participant wil complete a package of four questionnaires and the rheumatologist will assess disease activity. Participants assigned to VC-ERP will have their first two follow-up visits at an OTN site. There they will complete a package of four questionnaires, meet with the ERP for an assessment of disease activity, then connect with their rheumatologist by video conference. The final visit will take place in the rheumatologist's office, where the patient will complete a package of four questionnaires and the rheumatologist will assess disease activity.
5. Post-trial interview - 15 minute telephone interview that will be audio taped. Will take place no more than one month after final follow-up visit. Participants assigned to UC, will be asked the same questions as first interview. Participants assigned to VC-ERP, will be asked questions about their experience with the therapist and OTN during the study period

Significance: From perspective of people with stable, well-controlled IA, we will understand the barriers they perceive when travelling for rheumatology care far from their communities and whether this new model of care might help to mitigate some of that burden. This model already exists in Ontario and it's important to understand its value to people with stable IA and determine whether it is good use of an extended role practitioner's time.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years
* clinical diagnosis of inflammatory arthritis (i.e. rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis)
* inflammatory arthritis that is in remission or a low disease state as determined using a valid measure prior to study start
* travel to clinic ≥100 km round-trip
* able to read and write English
* willing/able to provide informed consent
* OHIP coverage.

Exclusion Criteria:

* Inflammatory arthritis that is neither in remission or in a low disease state as determined using a valid measure prior to study start
* complex rheumatic disease (i.e. lupus, vasculitis)
* travel to clinic <100 km round-trip
* children/youth < 18 years
* unable to read and write English
* unwilling/unable to provide informed consent
* no OHIP coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
European Quality of Life Questionnaire with 5 Dimensions and 5 Levels (EQ5D-5L) | 13 months
  Overall health:
  1. Rated in five dimensions as follows: Mobility from 1 (no problems) to 5 (unable to); Self-care from 1 (no problems) to 5 (unable to); Usual Activities from 1 (no problems) to 5 unable to); Pain/Discomfort from 1 (no pain) to 5 (extreme pain); Anxiety/Depression from 1 (not anxious/depressed) to 5 (extremely anxious/depressed)
  2. Rated on a visual analog scale from 0 (worst health you can imagine) to 100 (best health you can imagine).

SECONDARY OUTCOMES:
9-item Visit Satisfaction Questionnaire (VSQ9) | 13 months
  9 items on satisfaction with visit rated on a scale of 1 (poor) to 5 (excellent).
5-item Compliance Questionnaire Rheumatology | 13 months
  5 items on medication adherence rated on a scale of 1(strongly disagree) to 4 (strongly agree). Higher ratings indicate better adherence.
Health Assessment Questionnaire Disability Index (HAQ-DI) | 13 months
  Disability is evaluated by:
  1. rating 2 to 3 items in 8 dimensions (dressing & grooming, arising, eating, walking, hygiene, reach, grip, activities) from 0 (without any difficulty) to 3 (unable to do)
  2. indicating which aids, devices and assistance are needed
  3. Rating ability to carry out daily activities from 0 (completely) to 4 (not at all)
  4. Rating pain from 0 (no pain) to 100 (severe pain)
  5. rating overall health from 0 (very well) to 100 (very poor)
28-joint Disease Activity Score (DAS28- for rheumatoid arthritis) | 13 months
  Disease activity measure for IA patients with Rheumatoid Arthritis. Calculated with an algorithm using the following four items:
  1. Total number of swollen joints (out of a selected 28 joints specific to the disease)
  2. Total number of tender joints (out of a selected 28 joints specific to the disease)
  3. Global Health rated on a visual analog scale from 0 (well) to 100 (poor)
  4. Erythrocyte sedimentation rate (mm/hr) or C-reactive protein (mg/dl)
Disease Activity for Psoriatic Arthritis (DAPSA) | 13 months
  Disease Activity measure for IA patients with Psoriatic Arthritis Calculated as the sum of the following five items:
  1. Total number of swollen joints (out of a selected 66 joints specific to the disease)
  2. Total number of tender joints (out of a selected 66 joints specific to the disease)
  3. C-reactive protein (mg/dl)
  4. Disease activity rated on a visual analog scale from 0 (not active) to 10 (very active)
  5. Joint pain rated on a visual analog scale from 0 (none) to 10 (very severe)
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 13 months
  Disease activity measure for IA patients with Ankylosing Spondylitis. Calculated with an algorithm using the following five items:
  1. Back pain rated on a visual analog scale from 0 (none) to 10 (very severe)
  2. Peripheral pain/swelling rated on a visual analog scale from 0 (none) to 10 (very severe)
  3. Duration of morning stiffness rated on a visual analog scale from 0 (0 hrs) to 10 (2 hrs)
  4. Global health rated on a visual analog scale from 0 (well) to 10 (poor)
  5. Erythrocyte sedimentation rate (mm/hr) or C-reactive protein (mg/dl)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Dr. Henry Averns, Kingston, Ontario
  - Dr. Ashley Sterrett, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No